CLINICAL TRIAL: NCT01087294
Title: Administration of Anti-CD19-Chimeric-Antigen-Receptor-Transduced T Cells From the Original Transplant Donor to Patients With Recurrent or Persistent B-Cell Malignancies After Allogeneic Stem Cell Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 100054; 10-C-0054
Record Dates: First submitted 2010-03-13; First posted 2010-03-16 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-10-07

CONDITIONS: Leukemia, B-cell; Lymphoma, Hodgkins; Lymphoma, Non-hodgkins; Lymphoma, B-Cell
Keywords: CD19; Chimeric-Antigen-Receptor; Gene Therapy; Adoptive T Cell Therapy; Allogeneic Stem Cell Transplantation
MeSH Terms: conditions — Leukemia, B-Cell; Hodgkin Disease; Lymphoma, Non-Hodgkin; Lymphoma, B-Cell | interventions — Leukapheresis

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 1A/T cell Arm (closed) (Experimental): Dose escalation of CAR+ T cells based on the patients actual body-weight
  Interventions: Procedure: Allogeneic stem cell transplant; Biological: Anti-CD19-chimeric-antigen-receptor-transduced T cells
- 1B/T memory stem cell arm (Experimental): Dose Escalation with 5 dose levels of CAR+ T memory cells based on the patients actual body-weight
  Interventions: Procedure: Allogeneic stem cell transplant; Biological: Anti-CD19-chimeric-antigen-receptor-transduced T cells
- 2/Donor arm (Other): Leukapheresis
  Interventions: Procedure: Leukapheresis

INTERVENTIONS:
Procedure: Allogeneic stem cell transplant — Allogeneic stem cell transplant
  Arms: 1A/T cell Arm (closed); 1B/T memory stem cell arm
Biological: Anti-CD19-chimeric-antigen-receptor-transduced T cells — Patients receive T cells genetically engineered to express an anti-CD19 CAR. The cells are cultured in media containing IL-21, IL-7, and TWS119.
  TWS119 is a glycogen synthase 3 inhibitor
  Arms: 1A/T cell Arm (closed); 1B/T memory stem cell arm
Procedure: Leukapheresis — Donors will undergo leukapheresis
  Arms: 2/Donor arm

SUMMARY:
Background:

* Allogeneic hematopoietic stem cell transplantation (alloHSCT) is a procedure that transplants bone marrow cells (stem cells) from a matching donor into a recipient in order to allow the donor stem cells to produce cells that will attack the recipient s cancer cells. AlloHSCT is performed when chemotherapy, immunotherapy, or radiation therapy do not adequately control cancer growth. However, cancers that are not controlled by alloHSCT frequently become resistant to other standard treatment options.
* The outcomes of alloHSCT might be improved if certain kinds of white blood cells (T cells) could be manipulated so that they generate a more potent effect against the cancer cells. This effect can be augmented by genetically engineering donor T cells to specifically recognize cancerous cells in order to attack them. For this purpose, researchers are studying a specific kind of genetically engineered T cell known as the anti-CD19-CAR-transduced T cell. More research is needed to determine if this T cell will be an effective treatment for certain kinds of B cell cancer (such as non-Hodgkin s lymphoma and chronic lymphocytic leukemia) that has not been controlled with alloHSCT.

Objectives:

- To assess the safety and effectiveness of administering allogeneic anti-CD19-CAR-transduced T cells to patients with B-cell cancer that has not responded to alloHSCT.

Eligibility:

* Individuals between 18 and 75 years of age who have received allogeneic hematopoietic stem cell transplantation for a B cell cancer, but whose cancer has either not responded to or recurred after the transplant.
* Recipients must have the same stem cell donor from their previous procedure.

Design:

* Before the start of the study, all participants will be screened with a medical history and blood tests. Recipients will have tumor imaging scans, additional blood tests, and other tests as directed by the study doctors.
* Donor participants will undergo apheresis to provide white blood cells for researchers to use in the treatment.
* Recipients will have dose escalation to determine the most effective yet safe dose of anti-CD19 T cells. There will be six dose levels of anti-CD19 T cells. The first patients enrolled will have the smallest dose, and the dose will be increased when a level has been determined to be safe. .
* Recipients will be hospitalized for at least 9 days after receiving the cell infusion, and will need to come to clinic for follow-up visits 2, 4, 8, and 12 weeks after the infusion.
* Additional scans and frequent blood tests will be required for the first 3 months after the infusion, followed by less frequent visits over time.
* Recipients will be followed for a maximum of 15 years after receiving the infusion.

DETAILED DESCRIPTION:
Background:

Many patients with advanced B-cell malignancies that cannot be cured by chemotherapy and monoclonal antibodies have prolonged relapse-free survival after allogeneic hematopoietic stem cell transplantation (alloHSCT); however, a substantial fraction of patients with B-cell malignancies relapse following alloHSCT.

The first therapeutic maneuver attempted when patients without graft-versus-host disease (GVHD) relapse after alloHSCT is usually withdrawal of immunosuppressive drugs. If a remission does not occur after withdrawal of immunosuppression, patients are often treated with lymphocyte -DCI. Withdrawal of immunosuppression and DCI can lead to complete remissions in patients with B-cell malignancies that relapse after alloHSCT. Unfortunately, a substantial fraction of patients do not enter a complete remission after withdrawal of immunosuppression followed by DCI, and these therapies are often complicated by GVHD.

The outcomes of alloHSCT might be improved if T cells could be manipulated so that they generate a more potent graft-versus-malignancy (GVM) effect than unmanipulated T cells.

We hypothesize that the GVM effect against B-cell malignancies can be augmented by genetically engineering donor T cells to express receptors that specifically recognize antigens expressed by malignant B cells.

Chimeric antigen receptors (CARs) consist of an antigen recognition moiety combined with T-cell signaling domains. CARs are capable of activating T cells in an antigen-specific manner.

Expression of the CD19 antigen is limited to B cells and perhaps follicular dendritic cells. Most malignant B cells express CD19.

We have constructed a retroviral vector encoding an anti-CD19 CAR. Large numbers of T cells that have been transduced with this retroviral vector can be generated in vitro for clinical adoptive T cell therapy. These anti-CD19-CAR-transduced T cells specifically recognize a variety of CD19+ target cells and kill primary chronic lymphocytic leukemia (CLL) cells in vitro.

Primary Objective:

To assess the safety of administering allogeneic anti-CD19-CAR-transduced T cells to patients with B-cell malignancies that are persistent or relapsed after alloHSCT. The allogeneic anti-CD19-CAR-transduced T cells will be derived from the original allogeneic transplant donor.

Eligibility:

Patients with any CD19-expressing malignancy that is persistent or recurrent following successful engraftment after HLA-identical or >=9/10 matched sibling, 1-antigen mismatched sibling, or 9/10-matched unrelated donor (URD) alloHSCT and withdrawal of immunosuppression.

The same donor that provided cells for the alloHSCT must be willing and able to undergo leukapheresis so that cells can be obtained to prepare the anti-CD19-CAR-transduced T cells.

The recipient must have at most grade I acute GVHD or chronic GVHD with no organ site with a score exceeding 1, except for the skin, for which a score of 1 or 2 will be allowable. The recipient must not have received systemic immunosuppressive drugs given for graft versus host disease for at least 28 days at the time of study enrollment. Patients must be on a dose of corticosteroids of an equivalent of 5 mg/day or less of prednisone. Corticosteroid creams, ointments, and eye drops are allowed.

Design:

The alloHSCT donor will undergo leukapheresis.

Patients will undergo apheresis to obtain peripheral blood mononuclear cells. These cells will be processed to produce anti-CD19 CAR stem memory T cells (anti-CD19 CAR Tscm). This process involves sorting the cells and then culturing the cells in vitro for 9 days. During the 9-day culture period, the cells will be transduced with gammaretroviruses encoding the FMC63-28Z.

CAR recipients will be monitored for development of acute treatment-related toxicities for at least 9 days after cell infusion as inpatients. Dose-limiting toxicities (DLTs) will include severe acute GVHD and Grade 4 toxicities not associated with GVHD.

A maximum of 126 evaluable patients (donors plus recipients) will be treated.

Assessment of safety is a primary objective of this clinical trial. Safety will be defined as a lack of severe acute post-infusional toxicities and an incidence of GVHD that is not higher than historical rates of GVHD occurring after standard DCI.

Anti-CD19-CAR-transduced T-cell persistence in the peripheral blood will be measured at multiple time points from 1 week to 1 year after anti-CD19-CAR-transduced T cell infusion by flow cytometry.

To assess for an anti-malignancy effect of the infused cells, patients will be staged using standard staging systems.

ELIGIBILITY:
* INCLUSION CRITERIA:

Inclusion Criteria: Recipient

1. Recipients (patients with B-cell malignancy) must have received an HLA-identical or 9/10 matched sibling allogeneic hematopoietic stem cell transplant, or a greater than or equal to 9/10-matched unrelated donor (URD) alloHSCT for any CD19+ B-cell malignancy. Haploidentical donors will not be used in this protocol. Patients with any CD19+ B-cell malignancy that is persistent or relapsed after all of the following interventions are eligible:

   1. Donor engraftment after alloHSCT (>50% donor chimerism of the blood T cells or whole blood leukocytes or whole bone marrow).
   2. A trial of withdrawal of immunosuppressive therapy.

   NOTE: At least 28 days must have elapsed since the latest trial of withdraw of immunosuppression or DCI until the patient can be deemed to have persistent disease.
2. CD19 expression must be detected on the majority of the malignant cells by immunohistochemistry or by flow cytometry in the Laboratory of Pathology, CCR, NCI, NIH. Definition of which cells are malignant must be determined for each patient by the Laboratory of Pathology using techniques to demonstrate monoclonality such as kappa/lambda restriction (other techniques can be used to determine monoclonality at the discretion of the Laboratory of Pathology). The choice of whether to use flow cytometry or immuohistochemistry will be determined by what is the most easily available tissue sample in each patient. Immunohistochemistry will be used for lymph node biopsies and bone marrow biopsies. Flow cytometry will be used for peripheral blood, fine needle aspirate, and bone marrow aspirate samples.
3. Patients must be 18-75 years of age.
4. Performance status: ECOG less than or equal to 2
5. Either no evidence of GVHD or minimal clinical evidence of acute GVHD and chronic GVHD while off of systemic immunosuppressive therapy for at least 28 days. Minimal clinical evidence of acute GVHD is defined as grade 0 to I acute GVHD. Minimal evidence of chronic GVHD is defined as chronic GVHD with no organ site with a score exceeding 1, except for the skin, for which a score of 1 or 2 will be allowable (as defined by the 2005 NIH consensus project) or no chronic GVHD. Subjects with disease that is controlled to stage I acute GVHD or chronic GVHD meeting the above criteria with local therapy only, e.g., topical cutaneous steroids, will be eligible for enrollment.
6. Ability to give informed consent.
7. Prior Therapy: Therapy with monoclonal antibodies and/or chemotherapy must be stopped at least 14 days prior to anti-CD19 CAR-transduced T cell infusion, and recovery of treatment-associated toxicity to less than or equal to grade 2 is required prior to infusion of cells. For patients that have received prior DCI, the last dose must be at least 28 days prior to anti-CD19 CAR-transduced T cell administration. Note that patients can be enrolled on this study at any time after or during therapy, but at least 14 days must elapse from the time of prior monoclonal antibody administration or chemotherapy until anti-CD19 CAR-transduced T cells are infused, and at least 28 days must elapse from the time of withdraw of immunosuppression, or DCI, or other immunomodulatory therapies such as lenalidomide until anti-CD19 CAR-transduced T cells are infused. Systemic immunosuppression given for graft versus host disease must be stopped at least 28 days prior to protocol entry. There is no time restriction in regard to prior intrathecal chemotherapy provided there is complete recovery from any acute toxic effects of such.
8. Recipients of unrelated donor transplants from a National Marrow Donor Program (NMDP) Center must sign a release of information form to authorize NMDP transfer of information to the NIH.
9. Previous allogeneic donor must be willing and available to donate again.
10. Patients of childbearing or child-fathering potential must be willing use an effective method of contraception while being treated on this study and for 4 months after the last cell infusion.
11. Normal left ventricular function as evaluated by echocardiograph within 4 weeks of protocol therapy

Inclusion Criteria: Donor

1. Donors greater than or equal to 18 years of age must be the same individual whose cells were used as the source for the patient s original stem cell transplant.
2. Adequate venous access for peripheral leukapheresis, or consent to use a temporary central venous catheter for leukapheresis.
3. Donors must be HIV negative, hepatitis B surface antigen negative, and hepatitis C antibody negative.
4. Ability to give informed consent.
5. Donor selection will be in accordance with NIH/CC Department of Transfusion Medicine (DTM) criteria and, in the case of an unrelated donor from a Transplant Center, the National Marrow Donor Program (NMDP) standards. When a potentially eligible recipient of an unrelated donor product from an NMDP Center is identified, the recipient will complete an NMDP search transfer request to allow NIH NMDP staff to contact the NMDP Coordinating Center, who will, in turn, contact the donor s prior Donor Center. The NMDP Policy for Subsequent Donation Requests will be followed and the appropriate forms (Subsequent Donation Request form) and Therapeutic T Cell Collection Prescription will be submitted as required.

EXCLUSION CRITERIA:

Exclusion Criteria: Recipients

1. Active infection that is not responding to antimicrobial therapy.
2. Sero positive for HIV antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune -competence and thus are less responsive to the experimental treatment and more susceptible to its toxicities.)
3. Sero positive for hepatitis B antigen, positive hepatitis B tests can be further evaluated by confirmatory tests (HBV DNA), and if confirmatory tests are negative, the patient can be enrolled.
4. Sero positive for hepatitis C antibody unless antigen negative. If hepatitis C antibody test is positive, then patients must be tested for the presence of RNA by RT-PCR and be HCV RNA negative.
5. Active psychiatric disorder which may compromise compliance with the treatment protocol, or which does not allow for appropriate informed consent (as determined by Principal Investigator and/or his designee).
6. Pregnant or lactating. The effects of the immunosuppressive medications that could be required to treat GHVD are likely to be harmful to a fetus. The effects upon breast milk are also unknown and may be harmful to an infant.
7. Serum total bilirubin > 2.5 mg/dl, serum ALT and AST values greater than or equal to 2.5 times the upper limit of normal based on age-specific normal values. If the abnormal liver function is attributable to liver involvement by malignancy, patients may be eligible with serum total bilirubin up to 5.0 mg/dl, and serum ALT and AST values up to 5.0 times the upper limit of normal, provided the patient has no evidence of impending hepatic failure (encephalopathy or prothrombin time >2 time the upper limit of normal).
8. Serum creatinine greater than 1.6 mg/dL
9. Absolute neutrophil count of less than 1000 cells/ml unless low neutrophil count is thought to be due to malignancy in the bone marrow and malignancy is documented in the bone marrow.
10. Active cerebrospinal fluid involvement with malignancy or brain metastasis.
11. Platelet count less than 30,000/ml unless low platelet count is thought to be due to malignancy in the bone marrow and malignancy is documented in the bone marrow.
12. Hemoglobin less than 8.0 g/dL.
13. Receiving systemic corticosteroids including prednisone, dexamethasone or any other corticosteroid at doses of higher than 5 mg/day of prednisone within 28 days prior to anti-CD19-CAR-transduced T cell administration. Corticosteroid creams, ointments, and eye drops are allowed.
14. Blood blast percentage higher than 5%.

Exclusion Criteria: Donors

1. History of psychiatric disorder which may compromise compliance with this protocol or which does not allow for appropriate informed consent.
2. History of hypertension that is not controlled by medication, stroke, or severe heart disease (donors with symptomatic angina will be excluded). Donors with a history of coronary artery bypass grafting or angioplasty who are symptom free will receive a cardiology evaluation and be considered on a case-by-case basis.
3. Donors must not be pregnant.
4. Anemia (Hb < 11 gm/dl) or thrombocytopenia (platelets < 100,000 per ml). However, potential donors with Hb levels < 11 gm/dl that is due to iron deficiency will be eligible as long as the donor is initiated on iron replacement therapy. The NIH Clinical Center, Department of Transfusion Medicine/NMDP physicians will determine the appropriateness of individuals as donors.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2010-08-04 (Actual); Primary Completion 2024-03-08 (Actual); Study Completion 2024-04-02 (Actual)

PRIMARY OUTCOMES:
To assess the safety of allogeneic anti-CD19 CAR | 4-5 weeks after first dose
  List of adverse event frequency

SECONDARY OUTCOMES:
To measure the persistence of anti-CD19-CAR- transduced T cells in the blood of patients after infusion | Until the patient goes off-study for malignancy response assessment.
  Amount of anti-CD19-CAR- transduced T cells in the blood of patients after infusion.
To determine if administering anti-CD19-CAR-transduced T cells from the original transplant donor can cause regression of B-cell malignancies that are relapsed or persistent after alloHSCT | at progression
  Median amount of time subject survives without disease progression after treatment

CONTACTS AND LOCATIONS:
Overall Officials: James N Kochenderfer, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - National Marrow Donor Program, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.@@@@@@All collected IPD will be shared with collaborators under the terms of collaborative agreements.
Supporting Information: Study Protocol, SAP
Time Frame: Clinical data will be available during the study and indefinitely.@@@@@@Genomic data will be available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.@@@@@@Genomic data will be made available via dbGaP through requests to the data custodians.

REFERENCES:
- [Derived] Kochenderfer JN, Dudley ME, Carpenter RO, Kassim SH, Rose JJ, Telford WG, Hakim FT, Halverson DC, Fowler DH, Hardy NM, Mato AR, Hickstein DD, Gea-Banacloche JC, Pavletic SZ, Sportes C, Maric I, Feldman SA, Hansen BG, Wilder JS, Blacklock-Schuver B, Jena B, Bishop MR, Gress RE, Rosenberg SA. Donor-derived CD19-targeted T cells cause regression of malignancy persisting after allogeneic hematopoietic stem cell transplantation. Blood. 2013 Dec 12;122(25):4129-39. doi: 10.1182/blood-2013-08-519413. Epub 2013 Sep 20. PMID 24055823
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2010-C-0054.html